CLINICAL TRIAL: NCT04668703
Title: Prophylactic Effect of Conbercept Intravitreal Injection at the Conclusion of Cataract Surgery for Diabetic Macular Edema in Cataract Patients With Diabetic Retinopathy
Brief Title: Prophylactic Effect of Conbercept Intravitreal Injection at the Conclusion of Cataract Surgery for Diabetic Macular Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Yumeng Shi
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy; Cataract Diabetic
MeSH Terms: conditions — Diabetic Retinopathy | interventions — KH902 fusion protein

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined cataract surgery and intravitreal Conbercept injection (Experimental): Subjects will receive conbercept injections at a dose of 0.5 mg/eye at the conclusion of cataract surgery.
  Interventions: Procedure: Conbercept intravitreal injection
- cataract surgery alone (No Intervention): Subjects will undergo cataract surgery by phacoemulsification and intraocular lens implantation.

INTERVENTIONS:
Procedure: Conbercept intravitreal injection — intravitreal injection of 0.5 mg conbercept at the conclusion of cataract surgery
  Arms: combined cataract surgery and intravitreal Conbercept injection

SUMMARY:
Diabetic macular edema (DME) is an important cause of central vision impairment among people with diabetic retinopathy (DR), which can have a significant adverse effect on daily activities and quality of life. Diabetic patients with preexisting DME are at increased risk of worsening edema following cataract surgery. Previous studies also reported progression of DR after cataract surgery. Clinically significant DME is now classified into center-involved DME (CI-DME) and non center-involved DME (non-CI DME). Randomized clinical trials have established intravitreal antivascular endothelial growth factor (VEGF) therapy as first-line treatment for visual impairment from CI-DME and studies have addressed the influence of anti-VEGF therapy among patients with DME undergoing cataract surgery. However, for patients with non-CI DME before cataract surgery, whether anti-VEGF therapy is necessary at the end of surgery to prevent CI-DME is still clinically controversial. In order to evaluate the prophylactic effect of Conbercept (a recombinant fusion protein with high affinity to all VEGF isoforms and PIGF) intravitreal injection at the conclusion of cataract surgery for DME in patients with DR, the investigators will prospectively recruit 40 cataract patients with DR and non-CI DME and randomly assign these subjects into the study group (combined cataract surgery and intravitreal Conbercept injection, 20 cases) and the control group (cataract surgery alone, 20 cases). The primary outcomes include mean changes in central retinal thickness (CRT) and in diabetic retinopathy severity score (DRSS). The secondary outcomes include changes in best corrected visual acuity (BCVA), foveal avascular zone (FAZ), retinal vessel density (VD), the aqueous concentrations of VEGF, PIGF, interleukin- (IL-) 2, IL-5, IL-6, and IL-8.

ELIGIBILITY:
Inclusion Criteria:

* Patients sign informed consent, and are willing and able to comply with all the follow-ups
* Age ≥ 18 years , both genders
* Diagnosis of type 1 or type 2 diabetes mellitus
* Serum HbA1c ≤ 10%
* Patients with a diagnosis of DR (ETDRS 35-53) and cataract

Exclusion Criteria:

* CI-DME
* Any other ocular disorder in the study eye that may cause macular edema excluded the diabetic retinopathy
* History of allergic reaction to fluorescein, protein agents for diagnosis or therapy, or more than 2 drug or nondrug factors, or concomitant allergic diseases
* Received anti- VEGF treatment (including intravitreal injection or systematic application) within three months prior to enrollment
* History of panretinal laser photocoagulation (PRP) in the study eye 6 months prior to enrollment, or possibly need panretinal photocoagulation of the study eye during the study
* Intraocular conventional surgery within the past three months
* Traumatic cataract or congenital bilateral cataract in the study eye
* Active ocular or periocular infection in either eye
* Iris neovascularization in the study eye
* Uncontrolled glaucoma, or history of glaucoma surgery
* Aphakia in the study eye
* History of vitrectomy in the study eye
* The density of corneal endothelial cells is lower than 2000/mm2
* Patients with uncontrolled hyperglycemia, or Hemoglobin A1C (HbA1c) ≥10.0%, or under hemodialysis, or started insulin usage within the last 4 months, or expected to start insulin use for hyperglycemia control in the next 4 months
* Any surgical contraindications
* Uncontrolled Blood Pressure
* Myocardial infarction, heart failure, stroke, or transient ischemic attack within one month
* Renal Failure
* Pregnant or breast-feeding women
* Participation in another simultaneous medical investigator or trial
* Other situations where the researcher judges that the patient is not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
change in central retinal thickness (CRT) with optical coherence tomography (OCT) | Baseline, 1 month and 3 month after operation
  to compare the mean change from baseline of CRT between treatment group and control group at month 1 and 3
change in diabetic retinopathy severity score (DRSS) | Baseline, 1 month and 3 month after operation
  to compare the mean change from baseline of DRSS between treatment group and control group at month 1 and 3

SECONDARY OUTCOMES:
change in best corrected visual acuity (BCVA) | Baseline, 1 month and 3 month after operation
change in foveal avascular zone (FAZ) with optical coherence tomography angiography (OCTA) | Baseline, 1 month and 3 month after operation
change in retinal vessel density (VD) with optical coherence tomography angiography (OCTA) | Baseline, 1 month and 3 month after operation
change in the aqueous concentrations of VEGF, PIGF, interleukin- (IL-) 2, IL-5, IL-6, and IL-8 | Baseline, 1 week, 1 month and 3 month after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, MD, ph.D., Study Chair — Eye & ENT Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glassman AR, Wells JA 3rd, Josic K, Maguire MG, Antoszyk AN, Baker C, Beaulieu WT, Elman MJ, Jampol LM, Sun JK. Five-Year Outcomes after Initial Aflibercept, Bevacizumab, or Ranibizumab Treatment for Diabetic Macular Edema (Protocol T Extension Study). Ophthalmology. 2020 Sep;127(9):1201-1210. doi: 10.1016/j.ophtha.2020.03.021. Epub 2020 Mar 29. PMID 32402554
- [Background] Zhang J, Liang Y, Xie J, Li D, Hu Q, Li X, Zheng W, He R. Conbercept for patients with age-related macular degeneration: a systematic review. BMC Ophthalmol. 2018 Jun 15;18(1):142. doi: 10.1186/s12886-018-0807-1. PMID 29902977
- [Background] Relhan N, Flynn HW Jr. The Early Treatment Diabetic Retinopathy Study historical review and relevance to today's management of diabetic macular edema. Curr Opin Ophthalmol. 2017 May;28(3):205-212. doi: 10.1097/ICU.0000000000000362. PMID 28151747
- [Background] Peterson SR, Silva PA, Murtha TJ, Sun JK. Cataract Surgery in Patients with Diabetes: Management Strategies. Semin Ophthalmol. 2018;33(1):75-82. doi: 10.1080/08820538.2017.1353817. Epub 2017 Nov 16. PMID 29144826
- [Background] Grzybowski A, Kanclerz P, Huerva V, Ascaso FJ, Tuuminen R. Diabetes and Phacoemulsification Cataract Surgery: Difficulties, Risks and Potential Complications. J Clin Med. 2019 May 20;8(5):716. doi: 10.3390/jcm8050716. PMID 31137510
- [Background] Heier JS, Korobelnik JF, Brown DM, Schmidt-Erfurth U, Do DV, Midena E, Boyer DS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Vitti R, Berliner AJ, Zeitz O, Metzig C, Holz FG. Intravitreal Aflibercept for Diabetic Macular Edema: 148-Week Results from the VISTA and VIVID Studies. Ophthalmology. 2016 Nov;123(11):2376-2385. doi: 10.1016/j.ophtha.2016.07.032. Epub 2016 Sep 17. PMID 27651226
- [Background] Ip MS, Zhang J, Ehrlich JS. The Clinical Importance of Changes in Diabetic Retinopathy Severity Score. Ophthalmology. 2017 May;124(5):596-603. doi: 10.1016/j.ophtha.2017.01.003. Epub 2017 Mar 8. PMID 28284785
- [Background] Dhoot DS, Baker K, Saroj N, Vitti R, Berliner AJ, Metzig C, Thompson D, Singh RP. Baseline Factors Affecting Changes in Diabetic Retinopathy Severity Scale Score After Intravitreal Aflibercept or Laser for Diabetic Macular Edema: Post Hoc Analyses from VISTA and VIVID. Ophthalmology. 2018 Jan;125(1):51-56. doi: 10.1016/j.ophtha.2017.06.029. Epub 2017 Jul 29. PMID 28764888